CLINICAL TRIAL: NCT02493127
Title: The Effect of Priming of Questionnaire Content on Grip Strength in Patients With Hand and Upper Extremity Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015P000879
Record Dates: First submitted 2015-06-15; First posted 2015-07-09 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Hand and Upper Extremity Illness
MeSH Terms: interventions — Hand Strength

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard PCS (Experimental): Grip strength measurements and completes standard PCS
  Interventions: Other: Standard PCS; Other: Grip Strength
- Positive PCS (Experimental): Grip strength measurements and completes positively adjusted PCS
  Interventions: Other: Grip Strength; Other: Positively Adjusted PCS

INTERVENTIONS:
Other: Standard PCS — Subject completes the standard version of the PCS Questionnaire
  Arms: Standard PCS
Other: Grip Strength — Research Assistant takes Grip Strength Measurements
Other: Positively Adjusted PCS — Subject completes the positively-adjusted version of the PCS Questionnaire
  Arms: Positive PCS

SUMMARY:
Objectives:

To determine the association between priming and measurements of hand function such as grip strength

Primary null hypothesis:

There is no difference in grip strength (best of three attempts) as a percent of the opposite hand between patients that complete the standard Pain Catastrophizing Scale (PCS) compared to patients that complete the positively adjusted PCS.

Secondary null hypotheses:

There is no difference in grip strength (last of three attempts) as a percent of the opposite hand between patients that complete the standard PCS compared to patients that complete the positively adjusted PCS.

There is no difference in grip strength (best of three attempts) before and after completing the questionnaires between patients that complete the standard PCS compared to patients that complete the positively adjusted PCS.

DETAILED DESCRIPTION:
Priming affects all aspects of human behavior. Prior research by the investigators' group determined that completing a positively phrased version of the pain catastrophizing scale (PCS) primed patients to report less disability on average than completing the standard PCS. The influence of priming can be better understood by determining if it also affects direct measurements of hand function such as grip strength measures.

ELIGIBILITY:
Inclusion Criteria:

* All English-speaking adult patients visiting the Orthopaedic Hand and Upper Extremity Service

Exclusion Criteria:

* Unable to complete enrollment forms due to mental status or language problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Ring, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard PCS | Positive PCS
Started | 61 | 61
Completed | 60 | 60
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard PCS | Positive PCS | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (16) | 51 (16) | 53 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 26 | 61
  Male | 25 | 34 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 59 | 57 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 56 | 55 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
Grip Strength affected hand [Mean (Standard Deviation); unit: pounds] — Three grip strength measurements were recorded with the Dynamometer and the mean and maximum grip strength was calculated and reported.
  pounds
    Mean grip strength | 52 (24) | 62 (32) | 57 (28)
    Maximum grip strength | 56 (25) | 66 (32) | 60 (29)
Grip Strength of non-affected hand [Mean (Standard Deviation); unit: pounds] — Three grip strength measurements were recorded with the Dynamometer and the mean and maximum grip strength was calculated and reported.
  pounds
    Mean grip strength | 67 (28) | 75 (32) | 71 (30)
    Maximum grip strength | 72 (30) | 79 (33) | 76 (33)
Grip strength of both hands [Mean (Standard Deviation); unit: pounds] — Three grip strength measurements were recorded with the Dynamometer and the mean and maximum grip strength was calculated and reported.
  pounds
    Mean grip strength | 59 (23) | 68 (30) | 68 (30)
    Maximum grip strength | 73 (28) | 81 (33) | 78 (31)

OUTCOME MEASURES:

1. Primary Outcome: Pain Catastrophizing Scale (PCS)
Description: The pain catastrophizing scale is a 13-item scale to measure catastrophic thinking. The scale is from 0-4 and scores range from 0-52, a lower score indicates less catastrophic thinking about pain.
Time Frame: enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard Pain Catastrophizing Scale (PCS): Grip strength measurements and completes standard PCS
  Standard PCS: Subject completes the standard version of the PCS Questionnaire
  Grip Strength: Research Assistant takes Grip Strength Measurements
Arm/Group | Standard Pain Catastrophizing Scale (PCS)
Number analyzed (Participants) | 60
units on a scale | 8.2 (8.7)

2. Primary Outcome: Positive Pain Catastrophizing Scale (PCS)
Description: The positive pain catastrophizing scale (PCS) is a positively-phrased 13-item scale to measure catastrophic thinking. The scale is from 0-4 and scores range from 0-52, a higher score indicates less catastrophic thinking about pain.
Time Frame: enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive PCS
Number analyzed (Participants) | 60
units on a scale | 36.4 (9.8)

3. Primary Outcome: Difference in Grip Strength Measured With Dynamometer
Description: Difference in Grip strength of the non-affected hand after completing intervention. Each participant completed the grip strength measurement 3 times on the non-affected hand at enrollment (day 1). The results reported represent an increase or decrease in mean grip strength and maximum grip strength after completing the intervention.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Standard PCS | Positive PCS
Number analyzed (Participants) | 60 | 60
pounds
  Mean grip strength | 0.31 (5.3) | 2.2 (5.1)
  Maximum grip strength | -0.77 (7.2) | 1.8 (6.6)

4. Primary Outcome: Difference in Grip Strength Measured With Dynamometer
Description: Difference in Grip strength of the injured hand after completing intervention. Each participant completed the grip strength measurement 3 times on the injured hand at enrollment (day 1). The results reported represent an increase or decrease in mean grip strength and maximum grip strength after completing the intervention.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Standard PCS | Positive PCS
Number analyzed (Participants) | 60 | 60
pounds
  Mean grip strength | 1.3 (4.3) | 3.9 (6.2)
  Maximum grip strength | -0.17 (5.4) | 4.0 (7.3)

5. Primary Outcome: Difference in Grip Strength Measured With Dynamometer
Description: Difference in Grip strength of both hands after completing intervention. Each participant completed the grip strength measurement 3 times with both hands at enrollment (day 1). The results reported represent an increase or decrease in mean grip strength and maximum grip strength after completing the intervention.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Standard PCS | Positive PCS
Number analyzed (Participants) | 60 | 60
pounds
  Mean grip strength | 0.71 (4.1) | 3.1 (4.5)
  Maximum grip strength | -1.2 (6.9) | 2.7 (6.5)

ADVERSE EVENTS:
Arm/Group | Standard PCS | Positive PCS
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No